CLINICAL TRIAL: NCT01211964
Title: LEO 22811 - A Single Dose Bioavailability Study of Oral Solid Dosage Form Versus Oral Solution Including Fed Versus Fasted State in Healthy Male Subjects
Brief Title: LEO 22811 - Single Dose Bioavailability Study of Tablet Versus Oral Solution in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LEO 22811-S01; 2010-018388-41 (EudraCT Number)
Record Dates: First submitted 2010-09-23; First posted 2010-09-30 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2013-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LEO 22811 oral solution 1.5 mg (fasted state) (Experimental)
  Interventions: Drug: LEO 22811
- LEO 22811 single tablet 1.5 mg (fasted state) (Experimental)
  Interventions: Drug: LEO 22811
- LEO 22811 single tablet 1.5 (fed state) (Experimental)
  Interventions: Drug: LEO 22811

INTERVENTIONS:
Drug: LEO 22811 — Oral administration of solution and tablet.

SUMMARY:
The purpose of this phase 1 study is to determine the relative bioavailability and pharmacokinetics following single oral dose administration of LEO 22811 solution compared to LEO 22811 tablet in healthy male subjects as well as to determine the effect of food on the single oral dose pharmacokinetics of LEO 22811 tablet in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will prior to any study related activities, have given their written informed consent to participate in the study and to abide by the study restrictions
* Subjects will be Caucasian males between 18 and 55 years of age, with body mass index (BMI) between 18 and 32 kg/m2 both inclusive.
* Subjects will have a minimum weight of 50 kg
* Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations(congenital non-haemolytic hyperbilirubinaemia is acceptable)

Exclusion Criteria:

* Male subjects who are not willing to use appropriate contraception (such as condom)and for female partners; occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository) from the time of the first dose until 3 months after the final dosing occasion
* Subjects who have confirmed active/latent tuberculosis (TB)
* Subjects with an infectious illness within 3 days prior to dosing
* Subjects who have received any prescribed systemic or topical medication (including natural/herbal medicines) within 14 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration(with the exception of low to moderate use of vitamin/mineral supplements, however extreme vitamin use should be excluded) unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity), or a marketed drug within the past 3 months prior to the first dosing occasion.
* Subjects who have donated any blood, plasma or platelets in the month prior to screening or who have made donations on more than two occasions within the 12 months preceding the first dose administration
* Subjects with a significant history of drug allergy as determined by the Investigator
* Subjects who have any clinically significant allergic disease (excluding non-active hayfever) as determined by the Investigator
* Subjects who have a supine blood pressure and supine pulse rate at screening higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/40 mmHg and 45 bpm, respectively, confirmed by repeat
* Subjects who consume more than 28 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits)
* Subjects who smoke, or who have smoked within 3 months prior to first dose administration
* Subjects with, or with a history of, any clinically significant neurological, gastrointestinal,renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine,haematological, dermatological, autoimmunological or other major disorders as determined by the Investigator
* Subjects with a significant cardiac history (e.g. heart failure, hypokalemia, long QT syndrome) as determined by the investigator
* Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator
* Subjects who are known to have hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for HIV antibodies
* Subjects who, in the opinion of their General Practitioner (GP) or the investigator, should not participate in the study, including subjects suspected for whatever reason of not being able to comply with the requirements of the protocol
* Subject with serum levels of calcium, magnesium or potassium significantly outside the reference ranges. For subjects whose serum levels are not significantly outside these ranges, the physician may consult the sponsor with regards to approval for enrolment.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
AUC | 11 weeks
Tmax | 11 weeks
Cmax | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brooks, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No